CLINICAL TRIAL: NCT06508112
Title: Pleth Variability Index: A Potential New Marker for Predicting the Mortality of Pulmonary Embolism?
Brief Title: Pleth Variability Index in Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Teslime Eryavuz Şengül, Research assistant, Suleyman Demirel University
Other Study IDs: SuleymanDU-MED-TEŞ-01
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; Perfusion Index; Plethysmography; mortality
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed pulmonary embolism: Patients over the age of 18 who presented to the emergency department of a tertiary care hospital with complaints of cough, dyspnea, chest pain, tachycardia, hemoptysis, and syncope, and were diagnosed with pulmonary embolism (PE) confirmed by pulmonary computed tomographic angiography (CTPA), were included in our study. Informed consent was obtained from the patients who were stable and from the relatives of the patients who were unstable. Plethysmographic variability index (PVI) and Perfusion index (PI) levels were automatically obtained 2 minutes after the device was attached, using a probe placed on the index finger of the hand while the patient was lying supine. PI and PVI measurements and data were collected consecutively by the same individual. The measurements were taken using the Masimo Radical-7® Pulse CO-Oximeter, which is approved by the U.S. Food and Drug Administration.
  Interventions: Device: Masimo Radical-7® Pulse CO-Oximeter

INTERVENTIONS:
Device: Masimo Radical-7® Pulse CO-Oximeter — Masimo Radical-7® Pulse CO-Oximeter device was attached to the index finger of the patients in the supine position and photoplethysmographic perfusion index and plethysmographic variability index were measured noninvasively, rapidly and continuously.

SUMMARY:
Pulmonary embolism(PE) is a ventilation/perfusion disorder caused by obstruction of the pulmonary artery, usually by a thrombus. The Pleth Variability Index(PVI) is a continuous, noninvasive indicator of dynamic perfusion index changes in photoplethysmography that occur in at least one respiratory cycle. The aim of this study is to evaluate the prognostic and mortality indicator role of PVI in patients with PE, hypothesizing that PVI could serve as a valuable guide in this disease where perfusion impairment is fundamental.

Based on our study, we determined that PVI could be a non-invasive, rapid, and objective tool for predicting disease progression and mortality in PE patients in the emergency department. Our study is the first to evaluate the PVI in PE.

DETAILED DESCRIPTION:
Pulmonary embolism(PE) is a ventilation/perfusion disorder caused by obstruction of the pulmonary artery, usually by a thrombus. The Pleth Variability Index(PVI) is a continuous, noninvasive indicator of dynamic perfusion index(PI) changes in photoplethysmography that occur in at least one respiratory cycle. The aim of this study is to evaluate the prognostic and mortality indicator role of PVI in patients with PE, hypothesizing that PVI could serve as a valuable guide in this disease where perfusion impairment is fundamental.

In the emergency department, data were recorded for patients over 18 years of age diagnosed with pulmonary embolism, demographic data, risk scores and measurements. PVI and PI values were analyzed across different scoring systems, hospitalization statuses, and mortality groups. A survival analysis was conducted to evaluate the impact of PVI and PI on 1-year mortality in patients. The study was assessed with the STROBE checklist.

A total of 49 patients were included in this prospective, single-center study. The PVI value was significantly higher, whereas the PI value was significantly lower in the exitus group compared to the living group (p=0.027, p=0.011). The area under the curve values for PVI, pulmonary embolism severity index (PESI) score, and PI were determined to be 0.714, 0.820, and 0.745, respectively. It was observed that the negative predictive value of PESI was 100%, while the positive predictive value of PVI was the highest at 53.5%. In the. The mean survival time was significantly shorter for patients with PVI >40 and PI <1.9 (p=0.001, p=0.002). An increase in PVI was associated with a 4.04-fold increase in the risk of death (HR: 5.04, 95% CI: 1.50-16.92, p=0.009).

PVI can be considered a noninvasive, rapid, and objective tool for predicting the course and mortality of the disease in PE patients in the emergency department. Our study is the first to evaluate the PVI in PE.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old
* Diagnosis of pulmonary embolism

Exclusion Criteria:

* patients had asthma and chronic obstructive pulmonary disease exacerbation
* patients had acute decompensated heart failure
* patients were pregnant
* patient was under 18 years old

Ages: 18 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who presented to the emergency department of a tertiary care hospital between April 1, 2023, and March 31, 2024, with complaints of cough, dyspnea, chest pain, tachycardia, hemoptysis, and syncope, and were diagnosed with PE confirmed by pulmonary computed tomographic angiography (CTPA), were included in our study. Informed consent was obtained from the patients who were stable and from the relatives of the patients who were unstable.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pleth Variability Index: A Potential New Marker for Predicting the Mortality of Pulmonary Embolism? | 1 year
  PVI can be considered a noninvasive, rapid, and objective tool for predicting the course and mortality of the disease in PE patients in the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Teslime Eryavuz Şengül, M.D., Principal Investigator — suleyman demirel university faculty of medicine; Hamit H Armağan, assoc prof, Study Director — suleyman demirel university faculty of medicine; Furkan Ç Oğuzlar, asst prof, Study Chair — suleyman demirel university faculty of medicine
Locations (1):
- Suleyman Demirel University Faculty of Medicine, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No